CLINICAL TRIAL: NCT04456504
Title: HepB-CpG Series for Healthcare Workers Who Are Hepatitis B Vaccine Nonresponders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0631; A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison); Protocol Version 6/11/2020 (Other: UW Madison)
Record Dates: First submitted 2020-06-16; First posted 2020-07-02 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Healthcare Worker, Hepatitis B Vaccine, Nonresponder
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthcare worker (Experimental): Healthcare worker who has previously received at least 5 doses of hepatitis B vaccine with aluminum adjuvant (Recombivax B or Engerix B) and has an antibody to the hepatitis B surface antigen (antiHBs) that is less than 10 mIU/ml.
  Interventions: Biological: Recombinant hepatitis B vaccine with CpG adjuvant

INTERVENTIONS:
Biological: Recombinant hepatitis B vaccine with CpG adjuvant — Each participant will receive two doses of hepB-CpG separated by one month and blood draw to measure antibody to the hepatitis B surface antigen prior to dose 2 and one month after dose 2.

SUMMARY:
This study is being done to determine if healthcare workers who have previously failed to respond to hepatitis B vaccine series will respond to a hepatitis B with CpG adjuvant (hepB-CpG) (Heplisav-B)

DETAILED DESCRIPTION:
Study Intervention Each individual who has completed at least 5 doses hepB vaccine with aluminum adjuvant series but is anti-HBs negative will be contacted by EHS staff and invited to receive the hepB-CpG two dose series on a 0 and 1 month schedule. Antibody to the surface antigen will be measured after the first dose during the visit for the administration of the second dose. One month after completion of the series, each immunized individual will have another anti-HBs measured.

Total Number of Subjects Up to 130 individuals will be recruited and enrolled. Study Population Healthcare workers who have received at least 5 doses of hepatitis B vaccine with aluminum adjuvant and have antiHBs < 10mIU/ml.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Healthcare workers who have received at least 5 doses of hepatitis B vaccine with aluminum adjuvant and have antiHBs < 10mIU/ml
* Females of childbearing potential will be asked about the possibility of pregnancy as is the standard of care for immunization services. If a female indicates that she may be pregnant, study participation will be postponed until pregnancy is completed or the female reports that she is not pregnant.

Exclusion Criteria:

* Women who are pregnant or planning on becoming pregnant during the study
* Allergy to the vaccine or a component of the vaccine
* Not suitable for study participation due to other reasons, such as inability or unwillingness to comply with the study procedures, at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Russ RK, Vandehei HM, Golovkina MI, Mogallapalli H, Caldera F, Hayney MS. Hepatitis B-CpG Vaccine Series for Healthcare Workers Who Are Hepatitis B Vaccine Nonresponders. Clin Infect Dis. 2024 Aug 16;79(2):562-563. doi: 10.1093/cid/ciae320. PMID 38881506

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled from September 2020 to September 2023.
Period: Overall Study
Arm/Group | Healthcare Worker
Started | 49
Number of Participants Who Received First Dose | 49
Number of Participants Who Had Blood Draw After First Dose | 49
Number of Participants Who Received Second Dose | 48
Number of Participants Who Had Blood Draw After Second Dose | 47
Completed | 47
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthcare Worker
Number analyzed (Participants) | 49
Age, Customized [Count of Participants; unit: Participants]
  18-39 years old | 28
  40-59 years old | 16
  equal to or greater than 60 years old | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39
  Hispanic / Latinx | 3
  Black / African American | 2
  Asian | 3
  American Indian / Alaska Native | 2
Region of Enrollment [Number; unit: participants]
  United States | 49
Number of Prior Vaccine Doses [Count of Participants; unit: Participants]
  5 | 2
  6 | 44
  9 | 3
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 3
  Non-Smoker | 39
  Former Smoker | 7
Immunocompromised [Count of Participants; unit: Participants] — Immunocompromise was self-reported
  Participants
    Yes | 6
    No | 42
    Missing Data | 1
Diabetes [Count of Participants; unit: Participants]
  Yes | 4
  No | 45
Any Risk Factor [Count of Participants; unit: Participants] — Male, age >60 years, current smoker, immunocompromised, or diabetes; participants may have more than one risk factor
  Participants
    Yes | 31
    No | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Failed to Respond to 5 or More Doses of Hepatitis B Vaccine With Aluminum Adjuvant Who Respond to Hepatitis B Vaccine With CpG Adjuvant Series
Description: Response is defined as AntiHBs >10 mIU/ml following two doses of hepB-CpG
Time Frame: one month after dose 2 (up to 84 days on study)
Population: 1 participant dropped out of the study prior to the second dose, and 1 participant dropped out of the study prior to data collection post-second dose
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Worker
Number analyzed (Participants) | 47
Participants | 43

2. Secondary Outcome: Number of Participants Who Respond to a Single Dose of hepB-CpG
Description: Response is defined as AntiHBs >10 mIU/ml following a single dose of hepB-CpG
Time Frame: one month after dose 1 (up to 42 days on study)
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Worker
Number analyzed (Participants) | 49
Participants | 41

3. Secondary Outcome: Proportion of Participants Who Are Nonresponders With Each Risk Factor
Description: A multivariate model will be developed by measuring the proportion of participants who are nonresponders with each risk factor. Potential risk factors include including age, smoking status, sex, diabetes, immunosuppression.
Time Frame: one month after dose 2 (up to 84 days on study)
Population: Number of non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Worker
Number analyzed (Participants) | 4
Participants
  Male | 0
  Equal to or greater than 60 years old | 3
  Current Smoker | 0
  Immunocomprised | 1
  Diabetes | 0

ADVERSE EVENTS:
Time Frame: Adverse events data collected while participants are on study, up to 12 weeks
Description: Adverse Events are reported per dose, 49 participants for the first dose, and 47 of the 49 for the second dose as 2 participants were lost to follow up.
Groups:
- Healthcare Worker - Dose 1; Healthcare Worker - Dose 2: Healthcare worker who has previously received at least 5 doses of hepatitis B vaccine with aluminum adjuvant (Recombivax B or Engerix B) and has an antibody to the hepatitis B surface antigen (antiHBs) that is less than 10 mIU/ml.
  Recombinant hepatitis B vaccine with CpG adjuvant: Each participant will receive two doses of hepB-CpG separated by one month and blood draw to measure antibody to the hepatitis B surface antigen prior to dose 2 and one month after dose 2.
Arm/Group | Healthcare Worker - Dose 1 | Healthcare Worker - Dose 2
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 20/49 | 5/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthcare Worker - Dose 1 (N=49) | Healthcare Worker - Dose 2 (N=47)
Injection site soreness (Injury, poisoning and procedural complications) | 18 | 5
Chills (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT04456504/Prot_SAP_000.pdf